CLINICAL TRIAL: NCT01831843
Title: Effect of Breathing Circuits on Intraoperative Body Temperature
Acronym: BT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: php2
Record Dates: First submitted 2013-04-03; First posted 2013-04-15 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Brain Tumor
Keywords: core body temperature; humidity; circuit temperature
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group C (Placebo Comparator): non-heated, non-humidified conventional breathing circuit was used in group C patient
  Interventions: Device: Group C
- Group E (Experimental): breathing tube which apply humidity and heat (Evaqua™ Breathing Circuits manufactured by Fischer & Paykel)was used in group E patient
  Interventions: Device: Group E
- Group M (Experimental): Heated humid tube with a warming device (Mega Acer kit manufactured by Acemedical,Seoul Korea)was used in group M patient
  Interventions: Device: Group M

INTERVENTIONS:
Device: Group C — non-heated, non-humidified conventional breathing circuit was used in group C patient
  Other Names: conventional circuit
  Arms: Group C
Device: Group E — breathing tube which apply humidity and heat (Evaqua™ Breathing Circuits manufactured by Fischer & Paykel)was used in group E patient
  Other Names: Evaqua™ Breathing Circuits manufactured by Fischer & Paykel
  Arms: Group E
Device: Group M — Heated humid tube with a warming device (Mega Acer kit manufactured by Acemedical,Seoul Korea)was used in group M patient
  Other Names: Mega Acer kit manufactured by Acemedical,Seoul Korea
  Arms: Group M

SUMMARY:
To evaluate differences in intraoperative body temperature between heated huimid breathing circuit and conventional breathing circuit

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years,
* ASA I or II
* patients scheduled for craniotomy under general anesthesia

Exclusion Criteria:

* ASA III or IV
* Duration of anesthesia time less than 4 hours
* emergency operation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2013-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
trend of changes on body temperature | from the point of postintubation up to 5 hours
  Investigate differences on core body temperature among different kinds of circuit (heated-humid circuit, humid circuit, conventional circuit)

SECONDARY OUTCOMES:
total duration of airwarmer(Bair-Hurgger warming unit) using time | from the point of postintubation up to 5hours
  investigate the total duration of airwarmer using time

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim E, Lee SY, Lim YJ, Choi JY, Jeon YT, Hwang JW, Park HP. Effect of a new heated and humidified breathing circuit with a fluid-warming device on intraoperative core temperature: a prospective randomized study. J Anesth. 2015 Aug;29(4):499-507. doi: 10.1007/s00540-015-1994-z. Epub 2015 Mar 14. PMID 25771760